CLINICAL TRIAL: NCT02189148
Title: First-trimester Prediction of Preeclampsia and Other Placenta-mediated Pregnancy Complications
Brief Title: First-trimester Prediction of Preeclampsia
Acronym: PREDICTION
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Laval University (Other)
Responsible Party: Principal Investigator, Emmanuel Bujold, Principal Investigator, CHU de Quebec-Universite Laval
Other Study IDs: CIHR-MOP-133672; B14-05-2024 (Other: CER-CHU de Quebec)
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2018-07

CONDITIONS: Preeclampsia; Severe Preeclampsia; Fetal Growth Restriction; Preterm Birth
Keywords: Prediction; Preeclampsia; Preterm birth; Pregnancy; Placenta; Intra-uterine growth restriction; fetal growth restriction; Ultrasound; Doppler; Biomarkers; PAPP-A; Placental growth factor (PlGF)
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Each participant will :
  * give consent
  * provide a blood sample (10 ml)
  * be measured (weight and height for BMI calculation)
  * undergo a blood pressure measurement
  * have an ultrasound exam (uterine arteries Doppler, placental volume, thickness of the placenta)
  * answer to a short questionnaire (5 pages)

SUMMARY:
Preeclampsia is a complication of pregnancy related to adverse maternal and neonatal outcomes, including fetal growth restriction and perinatal death. Several measures are used or under investigation (low-dose aspirin, low-molecular weight heparin, calcium, folic acid, among others) for the prevention of preeclampsia. Unfortunately, most high-risk women who could benefit from those preventive measures are not identified until late in pregnancy. Recent evidences suggest that the investigators could identify women at risk of developing preeclampsia using a combination of serum and ultrasound biomarkers in the first-trimester of pregnancy. This screening test needs external validation. A first-trimester screening strategy will strengthen clinical research on preeclampsia and will contribute to the development of strategy combining the prediction and prevention of the disease and its related complications.

DETAILED DESCRIPTION:
Background: Preeclampsia (PE) is a placenta-mediated pregnancy complication related to adverse maternal and neonatal outcomes, including intra-uterine growth restriction (IUGR) and perinatal death. A growing body of evidence suggests that the preterm and severe forms of PE are associated with deep placentation disorders that occur early in gestation. Over the last decade, maternal characteristic and first-trimester biomarkers, including some that are already used for aneuploidy screening (PAPP-A) have been strongly related to the preterm and early forms of PE, suggesting that early prediction is possible. Preventive measures are actually recommended (low-dose aspirin; calcium) or under investigation (folic acid; low-molecular weight heparin; anti-oxidant) in high-risk women. However, only women with chronic disease or prior adverse pregnancy outcomes are eligible for these measures while most cases of PE occur in nulliparous women. Moreover, there are actually no clear guidelines for clinicians in Canada whose pregnant patients have one or several risk factors for preeclampsia (obesity, chronic hypertension, low PAPP-A, etc.). On the other hand, it has been suggested that prediction of PE, and particularly the most severe cases, is possible with high sensitivity and specificity by using a combination of anamnestic, biophysical, biochemical and ultrasonographic biomarkers using the web-based Fetal-Medicine Foundation (FMF) screening test. This suggests that a strategy of prediction and prevention of PE and other placenta-mediated complications is becoming possible for nulliparous women as well. However, certain major concerns must be addressed: 1) The FMF screening test has not been validated prospectively; 2) a controversy exists about the need and feasibility of Doppler ultrasound in the general population.

Objectives:

1. To validate the 11-13 week FMF screening test for early-onset PE and a composite of placenta-mediated outcomes (preterm PE, IUGR <3rd percentile, stillbirth); and
2. To compare the screening test with and without uterine artery (UtA) Doppler;
3. To explore the efficiency of new potential biomarkers (ADAM-12; Placental protein (PP) -13; placental and subplacental volume; placental vascularization) for prediction of PE in our population.

Methods: A multicenter prospective observational study of nulliparous women recruited between 11 3/7 - 13 6/7 weeks (maternal characteristics; BMI; Mean arterial pressure (MAP); PAPP-A; placental growth factor (PIGF); UtA Doppler…) and followed until delivery. Delivery and neonatal data will be collected through chart reviews. Detection rates for early-onset PE (primary outcome) and other adverse pregnancy outcomes will be measured using the 11-13 weeks FMF screening test with and without UtA Doppler results. A case-cohort study will be performed using stored serum samples and three-dimensional ultrasound volume acquired at the 11-13 weeks visit.

Feasibility and power calculation: We estimate a minimum incidence of early-onset PE of 0.7%. A minimum of 7,600 women will be necessary to demonstrate that the FMF screening test is at least 80% sensitive and 90% specific where it is expected that it will be 95% sensitive and 92% specific. We will have the power to detect an absolute difference of 15% in the detection rate between the different screening strategies (± Doppler). Recruitment will take 3.0 years. The overall study will take 5.0 years.

Expectations: First, our research will potentially provide a validated, highly sensitive and specific, and cheap tool to help clinicians' decision in the care of nulliparous women with risk factors for PE. In case of negative results, the clinician will have good evidence to reassure the patients facing abnormal maternal serum screening values. The validation of a first-trimester screening strategy will strengthen clinical research on PE providing new information on the natural evolution of the disease. Finally, this study will contribute to develop the optimal design for randomized trials aiming at the prevention of early-onset PE and other placenta-mediated complications of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 11 3/7 and 13 6/7 weeks;
* nulliparous women (no previous delivery ≥ 20 weeks).

Exclusion Criteria:

* pregnant women <18 years old at recruitment;
* multiple pregnancies;
* fetal congenital malformation;
* positive for HIV or hepatitis C or hepatitis B;
* negative fetal heart at recruitment;
* women planning a delivery outside the participating hospitals;
* women not able to provide an informed consent to the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nulliparous women who will deliver in one of the participating center:
  CHUL Hospital, Quebec city, QC Hôpital Saint-François-d'Assise, Quebec city, QC CHU Ste-Justine, Montreal, QC Southern Alberta Maternal Fetal Medicine Centre, Calgary, Alberta Sinai Health System, Mount Sinai Hospital, Toronto, Ontario
Sampling Method: Non-Probability Sample
Enrollment: 7554 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
early onset preeclampsia | diagnosed between 20 and 34 weeks of gestation
  Preeclampsia will be defined according to the Canadian Guidelines for Diagnosis, Evaluation, and Management of the Hypertensive Disorders of Pregnancy guidelines, as de novo hypertension with diastolic blood pressure >90 mmHg on two occasions at least four hours apart, after 20 weeks of pregnancy, associated with proteinuria ≥300 mg/24 h or at least '2 +' protein on urine dipstick or an adverse conditions

SECONDARY OUTCOMES:
Severe preeclampsia | between 20 and 42 weeks of gestation
  Severe Preeclampsia will be defined by the presence of at least one of the following adverse condition: 1) systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 110 mmHg after 4 h of bed rest, 2) proteinuria ≥ 5 g/24 h or at least '3 +' protein on urine dipstick, or 3) oliguria < 400 ml/24 h; 4) cerebral or visual disturbances; epigastric pain; pulmonary edema or cyanosis; thrombocytopenia <100,000mm
Fetal growth restriction | between 20 and 42 weeks of gestation
  Fetal growth restriction will be defined as a birth weight below the 10th centile (or below the 3rd centile for severe FGR) of Canadian reference growth charts.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bujold, MD, MSc, Principal Investigator — CHU de Québec; François Audibert, MD, MSc, Principal Investigator — St. Justine's Hospital
Locations (4):
- Canada (4):
  - South Alberta Maternal Fetal Medicine Centre, University of Calgary, Calgary, Alberta
  - Sinai Health System, Mount Sinai Hospital, Toronto, Ontario
  - CHU Ste-Justine, Montreal, Quebec
  - CHU de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerby P, Audibert F, Johnson JA, Okun N, Giguere Y, Forest JC, Chaillet N, Masse B, Wright D, Ghesquiere L, Bujold E. Prospective Validation of First-Trimester Screening for Preterm Preeclampsia in Nulliparous Women (PREDICTION Study). Hypertension. 2024 Jul;81(7):1574-1582. doi: 10.1161/HYPERTENSIONAHA.123.22584. Epub 2024 May 6. PMID 38708601
- See also: Prediction study at Centre de recherche du Centre Hospitalier Universitaire de Québec — http://www.crchudequebec.ulaval.ca/etudes/B14-05-2024.pdf